CLINICAL TRIAL: NCT04279899
Title: A Multicenter Observational Study of the Perinatal-neonatal Population With or With Risk of COVID-19 in China
Brief Title: The Investigation of the Neonates With or With Risk of COVID-19
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: CHFudanU_NNICU14
Record Dates: First submitted 2020-02-18; First posted 2020-02-21 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Neonatal Infection; Perinatal Problems; Infectious Disease
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Since December 2019, there has been an outbreak of novel coronavirus pneumonia in China. As of February 18, 2020, 72,530 cases confirmed with 2019 coronavirus disease(COVID-19) have been reported and 1,870 deaths were declared. Until now, cases of COVID-19 have been reported in 26 countries. This observational study aims to analysis the clinical features of neonates with COVID-19 and the neonates born to mother with COVID-19.

DETAILED DESCRIPTION:
Given that severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) spreads rapidly and is contagious to the general population, all the suspected or confirmed newborns will be admitted to the neonatal departments in designated hospitals of China. In this study, the diagnosis of neonatal SARS-CoV-2 infection is based on the criterion provided by National Health Commission and the Chinese perinatal-neonatal SARS-CoV-2 Committee. All samples will be treated as biohazardous material. SARS-CoV-2 will be tested in blood, cord blood, amniotic fluid, placenta, respiratory tract, stool, urine from mothers or neonates. The medical information questionnaires are classified into maternal and neonatal version, which include demographic details, epidemical history, clinical manifestations, tests collected time and results, imaging performed time and results and therapeutic data. Two researchers independently checked and recorded the data to ensure the accuracy of the data.

ELIGIBILITY:
Inclusion Criteria:

* The neonates with COVID-19,or neonates born by infected mothers

Exclusion Criteria:

* The neonates with major anomalies

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study participants will be recruited from all the designated hospitals in in 31 provinces/municipalities of the mainland of China during SARS-CoV-2 epidemic.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
The death of newborns with COVID-19 | The date of discharge，an average of 4 weeks after the admission
The SARS-CoV-2 infection of neonates born to mothers with COVID-19 | within 7days after the admission
  Neonates born to mothers with COVID-19 will be tested for SARS-CoV-2 after birth.Confirmed cases will meet the diagnosed criterion provided by National Health and Health Commission and the Chinese perinatal-neonatal SARS-CoV-2 Committee.

SECONDARY OUTCOMES:
The Chinese standardized Denver Developmental Screening Test (DDST) in neonates with or with risk of COVID-19 | Infants ( ≥35 weeks）are at 6 months after birth;Infants（< 35weeks） are at a corrected age of 6 months.
  The standardized DDST consists of 104 items and covers four areas of development: (a) personal/social, (b) fine motor/adaptive, (c) language, and (d) gross motor. In the present study, three trained professionals examined the children. The results of the DDST could be normal (no delays), suspect (2 or more caution items and/or 1 or more delays), abnormal (2 or more delays) or untestable (refusal of one or more items completely to the left of the age line or more than one item intersected by the age line in the 75-90% area). The children with suspect or abnormal results were retested 2 or 3 weeks later.
The small for gestational age newborns in the neonates born to mothers with COVID-19 | at birth
  The small for gestational age infant is defined as live-born infants weighting less than the 10th percentile for gestational age (22 weeks+0 day to 36 weeks+6days).
The preterm delivery of neonates born to mothers with COVID-19 | at birth
  The preterm infant is defined as the gestational age less than 37weeks+0day.The gestational age range is 22 weeks+0 day to 36 weeks+6days
The disease severity of neonates with COVID-19 | through study completion, estimated an average of 2 weeks
  Infants with SARS-CoV-2 infection are classified into asymptomatic, mild infection and severe infection, according to the expert consensus provided by the Chinese

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Maternal and Child Health Hospital of Hubei Province, Wuhan, Hubei
  - Children Hospital of Fudan University, Shanghai, Shanghai Municipality

REFERENCES:
- [Derived] Xiao T, Xia S, Zeng L, Lin G, Wei Q, Zhou W, Zhuang D, Chen X, Yi B, Li L, Mi H, Yin Z, Cheng X, Wang L, Hu X, Zhou W. A multicentre observational study on neonates exposed to SARS-CoV-2 in China: the Neo-SARS-CoV-2 Study protocol. BMJ Open. 2020 Jul 22;10(7):e038004. doi: 10.1136/bmjopen-2020-038004. PMID 32699166